CLINICAL TRIAL: NCT03356106
Title: Screening and Treatment of Obstructive Sleep Apnea in High-risk Pregnancy: A Multi-center Randomized Controlled Trial
Brief Title: Screening and Treatment of Obstructive Sleep Apnea in High-risk Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Visasiri Tantrakul, Dr., Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID11-58-12
Record Dates: First submitted 2017-09-26; First posted 2017-11-29 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Sleep Apnea, Obstructive; Pre-Eclampsia; Hypertension, Pregnancy-Induced
Keywords: Obstructive sleep apnea; Pre-Eclampsia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Experimental): Nocturnal administration of continuous positive airway pressure treatment (CPAP) until delivery
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Control (No Intervention): Usual antenatal care for high risk pregnancy

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — A non-invasive positive pressure device that is used for the treatment of obstructive sleep apnea by splinting the collapsed upper airway during sleep
  Arms: CPAP

SUMMARY:
This is an open-label multicenter randomized-controlled trial in 3 tertiary care hospitals including Ramathibodi Hospital, Phramongkutklao Hospital and Rajavithi Hospital. The study involved screening of obstructive sleep apnea in high risk pregnancy during 1st and 2nd trimesters. Randomization to either continuous positive airway pressure (CPAP) or usual antenatal care (ANC) until delivery will be done. Efficacy of CPAP on pregnancy outcome will be analysed.

DETAILED DESCRIPTION:
Screening for sleep disordered breathing (Respiratory disturbance index, RDI ≥ 5 events/hour) with type 2 sleep test will be performed in eligible subjects during early1st trimester (<16 weeks). Repeat sleep study will be done if the RDI in 1st trimester is less than 5. If the subjects meet the inclusion criteria without any of the exclusion criteria, randomization into either receiving CPAP treatment or usual ANC will be done. The pressure of CPAP machine is determined using autoCPAP machine algorithm at 90 percentile. Adjustment of CPAP machine is repeated at 24-28 week gestations. Subjects in both groups received standard usual care during ANC and outcomes were measured with similar case record forms.

ELIGIBILITY:
High risk pregnant women attending the antenatal care at the collaborated hospitals will be eligible for the study if they meet all following inclusion criteria.

Inclusion criteria (ALL criteria)

1. Singleton pregnant women age ≥ 18 years
2. Pregnant women attending the antenatal care and intending to deliver at one of the study hospitals with gestational age < 16 weeks
3. Thai nationality with ability to use Thai language proficiently both in spoken and written language.
4. Have been diagnosed as high-risk pregnancy by Obstetricians by having any of the following conditions

   1. Chronic hypertension prior to pregnancy
   2. Hypertension during pregnancy before 20 weeks gestation.
   3. Pre-eclampsia/gestational hypertension during recent pregnancy
   4. Obesity defined by pre-pregnancy body mass index (BMI) ≥ 27.5 kg/m2
   5. History of diabetes mellitus or gestational diabetes
   6. Having gestational diabetes or overt diabetes
5. Presence of snoring (either as frequent snoring ≥3 times/week or loud snoring) prior to or occurring during pregnancy OR respiratory disturbance index, RDI ≥ 5 events/hour by type 2 sleep testing at either point of testing during early pregnancy (0-16 GA week) or late pregnancy (GA 24-28week ).
6. Sign written informed consent

Exclusion Criteria:

1. Subjects' unwillingness to participate in the study at any time of the study.
2. Subject with significant medical conditions such as immunocompromised status, chronic infection (HIV infection, tuberculosis), chronic lung and cardiac conditions, chronic renal failure, thyroid disease, or neuromuscular disease.
3. Subjects with extremely severe obstructive sleep apnea (RDI ≥30) or with significant O2 desaturation <80% during sleep that might have potential benefit from the CPAP treatment.
4. Subject with known obstructive sleep apnea and currently on CPAP treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 340 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of blood pressure | During 24-28 weeks gestation
  Difference of daytime systolic and diastolic blood pressure between 2 groups (mmHg)
Measurement of blood pressure | During 32-34 weeks gestation
  Difference of daytime systolic and diastolic blood pressure between 2 groups (mmHg)
Measurement of blood pressure | During 24-28 weeks gestation
  Difference of daytime mean blood pressure between 2 groups (mmHg)
Measurement of blood pressure | During 32-34 weeks gestation
  Difference of daytime mean blood pressure between 2 groups(mmHg)
Measurement of blood pressure | During 18-20 weeks gestation
  Difference of daytime mean blood pressure between 2 groups (mmHg)
Measurement of blood pressure | During 18-20 weeks gestation
  Difference of daytime systolic and diastolic blood pressure between 2 groups (mmHg)

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure monitoring | measured twice during 24-28 week gestation, and 32-34 week gestation
  Using non-invasive technique from pulse transit time (SomnoTouch NIBP) (mmHg)
24-hour ambulatory blood pressure monitoring | measured twice during 32-34 week gestation
  Using non-invasive technique from pulse transit time (SomnoTouch NIBP) (mmHg)
Incidence of pregnancy induced hypertension (composite outcome1) | During pregnancy until delivery
  Incidence of hypertensive disorder of pregnancy
Incidence of hypertensive disorder of pregnancy or preterm labor or fetal growth restriction or emergency Cesarean section (composite outcome2) | During pregnancy until delivery
  Incidence of hypertensive disorder of pregnancy or preterm labor or fetal growth restriction or emergency Cesarean section
Incidence of preterm labor or fetal growth restriction or severe pre-eclampsia or eclampsia or death (composite outcome3) | During pregnancy until delivery
  Incidence of preterm labor or fetal growth restriction or severe pre-eclampsia or eclampsia or death
Fasting plasma glucose | during 24-28 weeks gestation
  Fasting plasma glucose (mg/dL)
Fasting plasma glucose | during 32-34 weeks gestation
  Fasting plasma glucose (mg/dL)
Oral glucose tolerance test (OGTT) | during 24-28 weeks gestation
  Oral Glucose Tolerance Test (OGTT) (mg/dL)
Fetal ultrasound results | During 24-28 weeks gestation
  Fetal growth (grams)
Fetal ultrasound results | During 32-34 weeks gestation
  Fetal growth (grams)
Fetal ultrasound results | During 18-20 weeks gestation
  Uterine Doppler arterial blood flow
Fetal ultrasound results | During 24-28 weeks gestation
  Uterine Doppler arterial blood flow
Fetal ultrasound results | During 32-34 weeks gestation
  Uterine Doppler arterial blood flow
Neonatal birthweight | at delivery
  Neonatal birthweight (grams)
APGAR score | at 1 minute and 5 minutes after birth
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form an acronym (Appearance, Pulse, Grimace, Activity, Respiration). Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
Neonatal length of stay in hospital | Through study completion up to 24 weeks
  Neonatal length of hospital stay (days) after birth until the newborn is discharged from the hospital
Neonatal ICU admission rate | Through study completion up to 24 weeks
  Neonatal ICU admission rate (%) after birth

CONTACTS AND LOCATIONS:
Overall Officials: Visasiri Tantrakul, MD, Principal Investigator — Ramathibodi Hospital Sleep Disorder Center, Pulmonary and Care division, Department of Medicine, Ramatibodi Hospital, Mahidol University, Thailand
Locations (3):
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No
For the first five years after the trial is concluded (upon acceptance of the primary manuscript for publication) the data will remain accessible only to the trial investigators for the purpose of additional analyses and publications. Thereafter other interested researchers may request in writing to the Steering Committee access to the data for the purpose of meta-analyses, with approval of a protocol and signed data access agreement via contacting the principle investigators of Division of Sleep Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Tantrakul V, Ingsathit A, Liamsombut S, Rattanasiri S, Kittivoravitkul P, Imsom-Somboon N, Lertpongpiroon S, Jantarasaengaram S, Somchit W, Suwansathit W, Pengjam J, Siriyotha S, Panburana P, Guilleminault C, Preutthipan A, Attia J, Thakkinstian A. Treatment of obstructive sleep apnea in high risk pregnancy: a multicenter randomized controlled trial. Respir Res. 2023 Jun 27;24(1):171. doi: 10.1186/s12931-023-02445-y. PMID 37370135

DOCUMENTS (1):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03356106/Prot_001.pdf